CLINICAL TRIAL: NCT06241677
Title: Intravenous Thrombolytic Therapy in Acute Ischemic Stroke Patients on Direct Oral Anticoagulants - a Prospective Multicenter Study
Brief Title: Intravenous Thrombolytic Therapy in Acute Ischemic Stroke Patients on DOAC
Acronym: DOAC-IVT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Pamela Youde Nethersole Eastern Hospital (Other); Queen Mary Hospital, Hong Kong (Other); Princess Margaret Hospital, Canada (Other); Tuen Mun Hospital (Other Government); The Queen Elizabeth Hospital (Other); United Christian Hospital (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB-2023-167-1
Record Dates: First submitted 2024-01-17; First posted 2024-02-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: CVA (Cerebrovascular Accident)
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator; Tenecteplase; TNK-tissue plasminogen activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVT group (Active Comparator): For patients enrolled into the IVT group from participating centers that allow IVT in patients with last DOAC intake 12-48 hours before presentation (PWH, QEH, QMH, UCH, TMH): Either alteplase (0.6 or 0.9mg/kg, maximum dosage 90mg, intravenous infusion) or tenecteplase (0.25mg/kg, maximum dosage 25mg, intravenous infusion) will be given at discretion of the treating physician.
  Interventions: Drug: alteplase or tenecteplase
- Control (No Intervention): For patients enrolled into the control group from participating centers that exclude eligible patients from IVT (PMH, PYNEH): no IVT will be given unless specific antidote can be administered before IVT.

INTERVENTIONS:
Drug: alteplase or tenecteplase — Either alteplase (0.6 or 0.9mg/kg, maximum dosage 90mg) or tenecteplase (0.25mg/kg, maximum dosage 25mg) will be given
  Other Names: tPA or TNK
  Arms: IVT group

SUMMARY:
Direct oral anticoagulants (DOAC) have emerged as safe and efficacious ischemic stroke prophylaxis for non-valvular atrial fibrillation (NVAF). All four DOACs - apixaban, dabigatran, edoxaban, rivaroxaban - were associated with lower risks of major bleeding compared to warfarin. Listed as core essential medicines by the World Health Organization, DOAC prescriptions have been surging worldwide. In Hong Kong, approximately 80,000 patients received DOACs from January 2009 through December 2022 according to the Hospital Authority registry.

The widespread DOAC usage had created DOAC-specific clinical dilemmas that lack evidence-based treatment despite twenty years of prescribing experience. Ischemic stroke despite DOAC (IS-DOAC), in particular, may occur in up to 6% of DOAC users annually. Due to the in vivo anticoagulation effect, there had been concerns of intracerebral bleeding (ICH) with intravenous thrombolytic therapy (IVT) for acute IS-DOAC. Under the current guideline recommendations, most acute IS-DOAC are contraindicated to IVT (see Intravenous thrombolytic therapy), which resulted in only a small proportion of acute ISDOAC patients being able to receive IVT even if presented early. Nonetheless, our group found that majority of patients had a DOAC level of <50ng/mL only 24 hours after DOAC cessation (see work done by us), a level deemed clinically negligible and safe for thrombolytic therapy. Together with evolving clinical evidence discussed below, IS-DOAC patients maybe unnecessarily barred from IVT, thus compromised functional recovery.

With robust pharmacokinetic and retrospective clinical evidence to support, it is hypothesized that IVT are safe in IS-DOAC patient. The investigators hereby propose a prospective multicenter study to determine the efficacy and safety of IVT in acute IS-DOAC.

DETAILED DESCRIPTION:
In this prospective cohort study, the investigators aim to recruit consecutive DOAC users with IS-DOAC who meet the inclusion criteria. The investigators aim to determine the safety and efficacy of IVT among DOAC patients with acute ischemic stroke. It is hypothesized that compared to a matched cohort of patients with acute IS-DOAC excluded from IVT, IVT in IS-DOAC patients with a last-DOAC-ingestion of 12-48 hours improves neurological outcomes with an acceptable safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke patients with a last-known-well to presentation time within 4.5 hours
2. Patients who took any doses of apixaban (2.5mg or 5mg twice daily), dabigatran (110mg or 150mg twice daily), edoxaban (30mg or 60mg daily) or rivaroxaban (15mg or 20mg daily) 12-48 hours before presentation
3. National Institute of Health Stroke Scale (NIHSS) ≥ 3
4. Alberta Stroke Programme Early CT (ASPECT) score ≥ 6
5. Pre-morbid modified Rankin Scale (mRS) ≤ 3
6. Patients aged ≥ 18 years old

Exclusion Criteria:

1. Initial CT brain showing intracranial haemorrhage
2. Contraindications to IVT according to current guideline recommendations [5], except for the use of DOAC within 12-48 hours
3. Patients with an estimated glomerular filtration rate of ≤ 30ml/min/1.73m2
4. Patients with bleeding propensities apart from the use of DOAC, e.g. platelet count of < 100x109/L
5. Patients with significant head injury immediately prior to presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2028-12-12 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Presence of symptomatic intracerebral hemorrhage (ICH) | up to 1 year
  As primary safety outcome. By the Heidelberg Bleeding Classification, the investigators shall categorize intracranial hemorrhages into HI1, HI2, PH1, PH2, and define symptomatic ICH as blood at any site in the brain with clinical deterioration (e.g. drowsiness and increased hemiparesis) or an increase in National Institute of Health Stroke Scale (NIHSS) score of ≥ 4 points (scores ranging from 0-42, higher scores indicating greater severity.)
Modified Rankin Scale (mRS) | 3 months after CVA
  To measure the degree of disability as a primary efficacy outcome, on the scale of 0-6: 0= no symptoms at all, 6=dead

SECONDARY OUTCOMES:
Presence of asymptomatic ICH | up to 1 year
  As seen from computer tomography (CT) and magnetic resonance imaging (MRI)
Presence of hemorrhagic transformation | up to 1 year
  As seen from computer tomography (CT) and magnetic resonance imaging (MRI)
Presence of malignant cerebral edema | up to 1 year
  As seen from computer tomography (CT) and magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventure Yiu Ming Ip, MB ChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No